CLINICAL TRIAL: NCT03978572
Title: The DART Study: Exercise Strategies to Improve Physical Function in Older Adults
Brief Title: Dual-benefits of Aerobic and Resistance Training
Acronym: DART
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Temporarily paused due to COVID-19 and expected to resume. Not of IRB approval
Sponsor: Ohio University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-F-55
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Sarcopenia; Aging; Disability Physical
Keywords: Exercise
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance Training (Active Comparator): 12 weeks of whole-body progressive resistance training, three days per week, lower-extremity focused (60% of exercises targeting lower extremities)
  Interventions: Behavioral: Resistance Training
- Moderate-intensity continuous cycling (Active Comparator): 12 weeks of progressive endurance cycling on a stationary bicycle at a target heart rate, three days per week.
  Interventions: Behavioral: Moderate-Intensity Continuous Cycling
- High-intensity interval cycling (Experimental): 12 weeks of progressive high-intensity interval cycling on a stationary bicycle, three days per week.
  Interventions: Behavioral: High-Intensity Interval Cycling

INTERVENTIONS:
Behavioral: Resistance Training — Exercise intervention designed to improve muscular strength and power
  Arms: Resistance Training
Behavioral: Moderate-Intensity Continuous Cycling — Exercise intervention designed to improve cardiorespiratory fitness and muscular endurance
  Arms: Moderate-intensity continuous cycling
Behavioral: High-Intensity Interval Cycling — Exercise intervention designed to improve cardiorespiratory fitness, muscular endurance, and muscular strength and power
  Arms: High-intensity interval cycling

SUMMARY:
This study evaluates the effect of three different exercise strategies on physical function in older adults. Participants will be randomly assigned to one of three exercise groups: resistance training, moderate-intensity continuous cycling on a stationary bicycle, and high-intensity interval training on a stationary bicycle.

DETAILED DESCRIPTION:
This project is confronting age-related physical disability by optimizing exercise strategies for older adults. Aerobic training is recommended to improve cardiorespiratory (heart and lung) function, while strength training is recommended for muscular function. These exercise effects are necessary for building healthier lives and reducing mortality and disability risk, but most older adults who do exercise typically only perform one type of exercise. In doing so they are missing a key component for healthy aging. This study will address whether stationary-cycling high-intensity interval training results in both cardiorespiratory and muscular improvements, and it will be the first controlled study comparing adaptations to high-intensity interval, aerobic, and strength training in sedentary older adults.

It is unclear whether the lack of muscular adaptations to traditional aerobic training is due to the low intensity/high volume model that is currently prescribed, and thus the central hypothesize of the study is that stationary-cycling high-intensity interval training can improve both cardiorespiratory and muscular function. To test this hypothesis, the investigators will measure heart, lung, and muscle function, as well as physical performance in sedentary older adults, before and after 12 weeks of supervised training using one of three exercise strategies; stationary-cycling high-intensity interval training, stationary-cycling moderate-intensity continuous training, or strength training. By comparing the outcomes across these three groups, the investigators will be able to confirm if short intervals of high-intensity exercise can elicit both cardiorespiratory and muscular benefits.

This work will demonstrate that older adults can improve their cardiovascular health and muscular strength with a single exercise strategy. Establishing in detail the cardiovascular and muscular benefits of this exercise can lead to the implementation of new and improved exercise guidelines for cardiovascular health and reduced physical disability in older adults. Incidentally, it will also provide a framework for future studies to investigate the importance of intensity in exercise. At the end of this study the investigators will be able to disseminate a new evidence-based exercise protocol that will address a significant barrier to healthy aging.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-75 years with no significant health issues or conditions that, in the investigator's opinion, would limit the subject's ability to complete the study per protocol or that would impact the capability to get an accurate measurement of study endpoints.
* Body mass index between 18.0 and 35 kg/m2.
* Willingness to maintain current diet and adhere to the intervention programs described for the study and willing to undergo all testing procedures.
* Able to read, understand, and complete study-related questionnaires
* Able to read and understand, and willing to sign the informed consent form (ICF).
* 6-minute walk distance of 450-725 meters for men and 400-675 meters for women.

Exclusion Criteria:

* Failure to provide informed consent.
* 6-minute walk distance below 450 meters or above 725 meters for men, below 400 meters or above 675 meters for women
* Any activities of daily living (ADL) disability (difficulty feeding, dressing, continence, bathing, toileting, and transferring).
* Lives in a nursing home or assisted living facility
* Known neuromuscular or neurological conditions affecting somatosensory or motor function or control (e.g., hemiplegia, multiple sclerosis, peripheral neuropathy, Parkinsons disease, Myasthenia Gravis, Ataxia, Apraxia, post-polio syndrome, mitochondrial myopathy, etc.).
* Unable to communicate because of severe hearing loss or speech disorder.
* Severe visual impairment, which would preclude completion of the assessments.
* Cancer requiring treatment currently or in the past 2 years (except primary non-melanoma skin cancer or in situ cervical cancer)
* Hospitalization (medical confinement for 24 hours), or immobilization, or major surgical procedure requiring general anesthesia within 12 weeks prior to screening, or any planned surgical procedures during the study period.
* Chronic or relapsing/remitting gastrointestinal disorders such as inflammatory bowel disease and irritable bowel syndrome.
* Known history of human immunodeficiency virus (HIV) antibody at screening.
* Use of systemic glucocorticoids.
* Any history of angina pectoris
* Any history of heart failure
* Any history of myocardial infarction
* Any coronary artery bypass graft or percutaneous coronary intervention
* Heart disease that limits exercise (valvular, congenital, ischaemic and hypertrophic cardiomyopathy)
* Complex ventricular arrhythmias or heart block
* Chronic obstructive pulmonary disease, cerebrovascular disease, or peripheral vascular disease
* Diabetes mellitus
* Severe neuropathy
* Mini-mental state exam score (MMSE) below 19
* Psychiatric conditions that warrant acute or chronic therapeutic intervention (e.g., major depressive disorder, bipolar disorder, panic disorder, schizophrenia) that in the investigators opinion may interfere with the conduct of study procedures
* Unable to undergo magnetic resonance imaging (MRI) (e. g. body containing any metallic medical devices or equipment, including heart pacemakers, metal prostheses, implants or surgical clips, any prior injury from shrapnel or grinding metal, exposure to metallic dusts, metallic shavings or having tattoos containing metallic dyes).
* Unable to reliably undergo exercise or strength tests described for this study.
* Participation in progressive resistance exercise 2 or more days/week for most weeks over the 24 weeks prior to screening, OR 150+ minutes of accumulated aerobic exercise each week for most weeks over the 24 weeks prior to screening.
* Current self-reported activity level that, in the investigator's opinion, is considered highly active for older adults
* Participation in any clinical trial within 12 weeks prior to screening.
* Limb amputation (except for toes) and/or any fracture within 24 weeks.
* Any disorder that will not allow completion of the motions required for resistance or aerobic exercise
* Conditions (such as myasthenia gravis, myositis, muscular dystrophy or myopathy, including drug-induced myopathy) leading to muscle loss, muscle weakness, muscle cramps or myalgia.
* Acute viral or bacterial upper or lower respiratory infection at screening
* Abnormal or uncontrolled blood pressure (BP) at the screening visit defined as BP > 170/100 mmHg. If taking anti-hypertensive medication, have to be on stable doses of medication for more than 3 months.
* Current or recent history (within 1 year of screen) of heavy alcohol consumption or drug abuse that in the investigators opinion may interfere with the conduct of study procedures.
* Reports being pregnant, lactating, or that they anticipate becoming pregnant in the next 3-months. If a woman becomes pregnant while on study protocol they will be withdrawn from the study

Prohibited Medications: Medications that, in the PIs opinion, would confound study integrity by interacting with study outcomes. For instance:

* Anti-obesity drugs, nutraceuticals, and dietary supplements that may affect body mass and body composition.
* Any drug or supplement known to influence muscle mass or performance including but not limited to anabolic steroids, insulin-like growth factor 1 (IGF-1), growth hormone (GH), replacement androgen therapy, anti-androgen therapy.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximal Oxygen Consumption | Change from baseline at 12 weeks
  The primary endpoint is maximal oxygen consumption measured by both relative and absolute changes in maximal oxygen consumption obtained during a graded exercise test on a cycle ergometer.
Knee extensor isokinetic power | Change from baseline at 12 weeks
  Maximal muscle power (maximal torque in foot-pounds) of the quadriceps using an isokinetic dynamometer

SECONDARY OUTCOMES:
Knee extensor isometric force production | Change from baseline at 12 weeks
  Maximal muscle strength of the quadriceps (in foot-pounds) as measured by an isometric dynamometer
Knee extensor isokinetic endurance | Change from baseline at 12 weeks
  Total power output (cumulative torque in foot-pounds) produced from 120 consecutive maximal knee extensions using an isokinetic dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Clark, PhD, Study Chair — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tavoian D, Russ DW, Law TD, Simon JE, Chase PJ, Guseman EH, Clark BC. A Randomized Clinical Trial Comparing Three Different Exercise Strategies for Optimizing Aerobic Capacity and Skeletal Muscle Performance in Older Adults: Protocol for the DART Study. Front Med (Lausanne). 2019 Oct 22;6:236. doi: 10.3389/fmed.2019.00236. eCollection 2019. PMID 31750307